CLINICAL TRIAL: NCT01773044
Title: Pain on Injection of Propofol: a Comparison of Lidocaine and Alkalinized Lidocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, department of anesthesiology, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ulkü_1
Record Dates: First submitted 2012-12-20; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Pain on Injection of Propofol,Lidocaine, Alkalinized Lidocaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- alkalinized lidocaine & lidocaine (Active Comparator)
  Interventions: Drug: alkalinized lidocaine; Drug: Lidocaine
- alkalinized lidocaine &Placebo (Active Comparator)
  Interventions: Drug: alkalinized lidocaine; Drug: Placebo (for alcalinized lidocaine)

INTERVENTIONS:
Drug: alkalinized lidocaine — recevied 0.05 mL/kg lidocaine with bicarbonate ( % 2 lidocaine 5 mL + 1 mL %8,4 NaHCO3+ 4 mL SF)
Drug: Lidocaine — 0.05 mL/kg lidocaine (% 2 lidocaine 5 mL + 5 mL SF),
  Arms: alkalinized lidocaine & lidocaine
Drug: Placebo (for alcalinized lidocaine)
  Arms: alkalinized lidocaine &Placebo

SUMMARY:
Aim: The aim of this study was to compare the efficacy of pretreatment 0.5 mg/kg lidocaine and 0.5 mg/kg alkalinized lidocaine for prevention of propofol induced pain.

Methods: In this double-blind, placebo controlled study, 300 adults patients ASA I or II, scheduled to undergo elective surgery, were randomly assigned into three groups of 100 each. Group L, recevied 0.05 mL/kg lidocaine (% 2 lidocaine 5 mL + 5 mL SF), Group A, 0.05 mL/kg lidocaine with bicarbonate ( % 2 lidocaine 5 mL + 1 mL %8,4 NaHCO3+ 4 mL SF) and control group received isotonic saline pretreatment in the dorsum of the hand, followed by propofol 30 sec later. A blinded researcher assessed the patient's pain level via a four-point scale.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective surgery

Exclusion Criteria:

* allergy to the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pain on injection of propofol | 5 th minutes after propofol injection

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu university medicine faculty, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Borazan H, Erdem TB, Kececioglu M, Otelcioglu S. Prevention of pain on injection of propofol: a comparison of lidocaine with different doses of paracetamol. Eur J Anaesthesiol. 2010 Mar;27(3):253-7. doi: 10.1097/EJA.0b013e328330eca2. PMID 19696679